CLINICAL TRIAL: NCT03267914
Title: Impact of Compliance With Fluoride Use on Caries Incidence After Cancer Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: A.T. Still University of Health Sciences (Other)
Responsible Party: Principal Investigator, Seena Patel, Dentist, Associate Director of Oral Medicine and Assistant Professor, A.T. Still University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-005
Record Dates: First submitted 2017-08-14; First posted 2017-08-31 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Dental Caries; Oral Cavity Cancer; Oral Complications of Chemotherapy and Head/Neck Radiation
MeSH Terms: conditions — Dental Caries; Mouth Neoplasms | interventions — traY protein, E coli; Toothbrushing

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to receive fluoride therapy with either custom trays (Tray group) or by application with a toothbrush (Brush group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tray group (Experimental): Control intervention Patients will use the custom-made tray to apply the fluoride locally to the teeth and wear for 5 minutes each day.
  Interventions: Other: Tray
- Brush group (Active Comparator): Patients will brush with the fluoride for 2 minutes each day.
  Interventions: Other: Brush

INTERVENTIONS:
Other: Tray — Control intervention Patients will use the custom-made tray to apply the fluoride locally to the teeth and wear for 5 minutes each day.
  Arms: Tray group
Other: Brush — Patients will brush with the fluoride for 2 minutes each day.
  Arms: Brush group

SUMMARY:
Approximately 40 people will participate in this study. This study will compare two different methods of fluoride application. Both methods are currently used in dental practice and both have been shown to be effective. If the participant chooses to participate in this study, participant will be asked to either wear a small tray that has been custom made to fit into the mouth into which fluoride is placed and worn for 5 minutes at bedtime, or participant will be asked to brush fluoride onto the teeth for 2 minutes at bedtime. Participant will be randomly assigned to use one of these methods of fluoride application: participant will not be allowed to choose which method of application you prefer. Participant will be asked to use fluoride every night while enrolled in the study. The fluoride that is used in the study is approved by the United States Food and Drug Administration and is commercially available with a prescription. After the study is over, participant will need to continue to use fluoride every night for life to help reduce the risk for dental cavities in the future.

During the study, participant will receive a dental examination every 3 months for a total of 4 study visits over the period of 1 year. This visit will consist of a dental examination to identify any new cavities and instructions for fluoride use. Participant will also be asked to complete a written log to document daily fluoride use and to give feedback about compliance with fluoride use.

DETAILED DESCRIPTION:
This research proposal is unique in that it compares two different methods of applying neutral sodium fluoride to prevent dental caries and improve compliance in this at-risk population. Given that compliance with use of fluoride trays has historically been poor, there is controversy as to which application method is best. Further, the optimal dosage regimen is unknown. Clarification is needed to support best practices.

Data from the proposed study will help to identify an effective and tolerated form of fluoride delivery in patients undergoing head and neck radiation therapy. If our hypotheses are supported, additional studies will be undertaken with a larger sample size, and expanded to include patients with head and neck cancers treated with chemotherapy or a combination of cancer therapies.

All patients will undergo an initial dental visit, which will consist of medical consultation with the patient's oncologist and standard dental and radiographic examinations. Patients will return to have existing dental disease treated (eg. caries, gingival disease, extractions). When treatment is complete, they will be invited to participate in the study. The Screening Form will be used to confirm eligibility.

Study Visit #1 (Baseline) After obtaining consent, subjects will be randomly assigned to receive fluoride therapy with either custom trays (Tray group) or by application with a toothbrush (Brush group). Each subject will undergo a basic dental examination for identification of new carious lesions. Visit #1 is the baseline, with a new caries score of zero. Photographs will be taken of the subject's mouth and instructions for fluoride therapy will be given.

Tray group: The subject will have custom vinyl vacuform fluoride trays made using an in-house laboratory. They will be instructed to apply a "ribbon" of fluoride gel into each tray, and then to wear each tray for 5 minutes, one tray at a time, after which the subject will expectorate any remaining fluoride from the mouth.

Brush group: The subject will be instructed to apply a "ribbon" of fluoride gel onto the toothbrush provided (Colgate Wave Sensitive) and to brush with the fluoride for 2 minutes at bedtime.

Both groups: The subject may not rinse, eat, or drink for 30 minutes after the fluoride treatment.

All subjects will be instructed to perform their fluoride therapy at bedtime and to document the date and time of treatment on the Monthly Fluoride Log. All subjects will be provided with 1.1% neutral sodium fluoride (PreviDent®) gel for the duration of the study. All subjects will be instructed to return their monthly fluoride logs and any remaining fluoride at each study visit.

Subjects will return for a follow-up examination at 3, 6, 9, and 12 months from the first study visit. At each visit, the following procedures will be conducted:

* Update medical history
* Take photographs
* Conduct examination for caries
* Assess compliance with fluoride therapy
* Collect fluoride log for previous 3 months
* Dispense new fluoride log
* Collect and weigh returned fluoride tube
* Weigh and dispense new fluoride tube
* Dispense new toothbrush (Brush group only)

Subjects will be scheduled to immediately return to have any new carious lesions filled.

To evaluate compliance, subjects will be asked about their fluoride use according to standard methods utilized by other experts in the field. High compliance is defined as daily use; low compliance is defined as two to three times per week; not compliant is defined as less than two times per week.

To evaluate caries incidence, the number of surfaces per tooth on which new caries appear will be documented on the Caries Assessment Form. Caries will be scored using the International Caries Classification and Management System criteria for clinical research. Surfaces will be scored as either I (no obvious decay) or II (obvious decay). Bitewing radiographs and periapical films (as needed) will be taken at 6 and 12 months after the initial examination visit.

Descriptive statistics, including means (standard deviations) or counts (percentages), as appropriate, will be used to summarize baseline demographic and clinical characteristics of the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Diagnosis of cancer in the head and neck region
* Field of radiation must include the parotid gland(s) and/or submandibular gland region
* Able to speak English
* Able to provide consent
* Able to return for all study visits

Exclusion Criteria:

* Previous/current use of prescription strength fluoride
* Previous history of radiation to the head and neck region
* Presence of autoimmune disease(s)
* Currently pregnant
* Currently edentulous or will become edentulous prior to beginning radiation therapy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
Fluoride use compliance | 3 months
  To evaluate compliance, subjects will be asked about their fluoride use according to methods described by Epstein et al. (1996). High compliance is defined as daily use; low compliance is defined as two to three times per week; not compliant is defined as less than two times per week.
Fluoride use compliance | 6 months
  To evaluate compliance, subjects will be asked about their fluoride use according to methods described by Epstein et al. (1996). High compliance is defined as daily use; low compliance is defined as two to three times per week; not compliant is defined as less than two times per week.
Fluoride use compliance | 9 months
  To evaluate compliance, subjects will be asked about their fluoride use according to methods described by Epstein et al. (1996). High compliance is defined as daily use; low compliance is defined as two to three times per week; not compliant is defined as less than two times per week.
Fluoride use compliance | 12 months
  To evaluate compliance, subjects will be asked about their fluoride use according to methods described by Epstein et al. (1996). High compliance is defined as daily use; low compliance is defined as two to three times per week; not compliant is defined as less than two times per week.

SECONDARY OUTCOMES:
Dental caries incidence assessed at 4 time points | 3 months
  To evaluate caries incidence clinically, the number of surfaces per tooth on which new caries appear will be documented on the Caries Assessment Form. Caries will be scored using the International Caries Classification and Management System criteria for clinical research. Surfaces will be scored as either I (no obvious decay) or II (obvious decay).
Dental caries incidence assessed clinically at 4 time points | 6 months
  To evaluate caries incidence clinically, the number of surfaces per tooth on which new caries appear will be documented on the Caries Assessment Form. Caries will be scored using the International Caries Classification and Management System criteria for clinical research. Surfaces will be scored as either I (no obvious decay) or II (obvious decay).
Dental caries incidence assessed at 4 time points | 9 months
  To evaluate caries incidence clinically, the number of surfaces per tooth on which new caries appear will be documented on the Caries Assessment Form. Caries will be scored using the International Caries Classification and Management System criteria for clinical research. Surfaces will be scored as either I (no obvious decay) or II (obvious decay).
Dental caries incidence assessed at 4 time points | 12 months
  To evaluate caries incidence clinically, the number of surfaces per tooth on which new caries appear will be documented on the Caries Assessment Form. Caries will be scored using the International Caries Classification and Management System criteria for clinical research. Surfaces will be scored as either I (no obvious decay) or II (obvious decay).

OTHER OUTCOMES:
Dental caries incidence assessed radiographically at 2 time points | 6 months
  To evaluate caries incidence radiographically, bitewing radiographs and periapical films (as needed) will be taken at 6 and 12 months after the initial examination visit.
Dental caries incidence assessed radiographically at 2 time points | 12 months
  To evaluate caries incidence radiographically, bitewing radiographs and periapical films (as needed) will be taken at 6 and 12 months after the initial examination visit.

CONTACTS AND LOCATIONS:
Overall Officials: Seena Patel, DMD, MPH, Principal Investigator — A.T. Still University, Arizona School of Dentistry & Oral Health
Locations (1):
- A.T. Still University, Arizona School of Dentistry & Oral Health, Mesa, Arizona, United States

IPD SHARING:
Plan to Share IPD: No